CLINICAL TRIAL: NCT07240012
Title: Automated Insulin Delivery Versus Usual Insulin Treatment Modality Before and During Pregnancy in Women With Type 1 Diabetes
Acronym: AID-DM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The Novo Nordic Foundation (Other); mylife Diabetes Care AG (Industry); Abbott (Industry)
Responsible Party: Principal Investigator, Lene Ringholm, Chief physician, PhD, Associate Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3080181
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-11

CONDITIONS: Diabete Type 1; Pregnancy Complications
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Automated closed-loop insulin delivery (AID) (Experimental)
  Interventions: Device: Automated closed-loop insulin delivery
- Usual insulin treatment modality (No Intervention)

INTERVENTIONS:
Device: Automated closed-loop insulin delivery — Automated closed-loop insulin delivery and The mylife CamAPS FX algorithm combined with CGM
  Arms: Automated closed-loop insulin delivery (AID)

SUMMARY:
A national multi-center open-label randomized controlled trial that investigates whether the use of the automated insulin delivery system CamAPS FX initiated during pregnancy planning or in early pregnancy improves maternal time in glycemic targets and fetal growth in women with type 1 diabetes compared to usual insulin treatment modality combined with Continuous Glucose Monitoring.

DETAILED DESCRIPTION:
This is a national multi-center open-label randomized controlled trial investigating whether the use of the automated insulin delivery system CamAPS FX initiated during pregnancy planning or in early pregnancy (<14 completed weeks) improves maternal glycemic control in women with type 1 diabetes during pregnancy, delivery and post-delivery and leads to more appropriate fetal growth compared to usual insulin treatment modality (multiple day injections or insulin pump) combined with continuous glucose monitoring.

Women planning pregnancy will initiate the automated insulin delivery system CamAPS FX or continue usual insulin treatment modality combined with a compatible continuous glucose monitoring, as per randomisation allocation before conception and throughout pregnancy until one month post-delivery or for up to 52 weeks if not becoming pregnant. Women who become pregnant during the 52-week study period will be referred to their local center for pregnant women with diabetes and followed during pregnancy until one month post-delivery. Women who do not become pregnant during the 52-week study period will leave the study and continue usual diabetes care at their usual diabetes center.

Women who are pregnant at randomisation will initiate the automated insulin delivery system CamAPS FX or continue usual insulin treatment modality combined with a compatible continuous glucose monitoring as per randomisation allocation, throughout the pregnancy period until one month post-delivery.

ELIGIBILITY:
Inclusion criteria during pregnancy planning

* Women, age 18-45 years
* Duration of type 1 diabetes ≥ 12 months
* Women who are not pregnant confirmed by a negative pregnancy test on the day of randomization
* Planning pregnancy within 52 weeks

Inclusion during pregnancy:

* Women, age 18-45 years
* Duration of type 1 diabetes ≥ 12 months
* Pregnant with an intrauterine singleton living fetus confirmed by an ultrasound scan between 8+0 and 13+6 gestational weeks
* Accepting participation in the DDBR2 study during pregnancy, delivery and until one month after delivery

Exclusion criteria during pregnancy planning and during pregnancy:

* No proficiency in Danish to understand oral and written information
* Severe mental or psychiatric barriers or concurrent disease on the decision of the principal investigator

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 305 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Time in range | From first day of last menstrual cycle (planning pregnancy) or randomization (early pregnancy) until delivery.
  The between group difference in time in range in pregnancy (3.5-7.8 mmol/L) between intervention and controls
Neonatal outcome: Birthweight | At delivery
  Offspring birthweight standard deviation score adjusted for gestational age and infant gender.

SECONDARY OUTCOMES:
Continuous glucose monitoring data | From randomisation during pregnancy planning until delivery or leaving study after 52 weeks (randomized during pregnancy planning) or from randomization in early pregnancy to delivery
  Mean sensor glucose, mean sensor glucose coefficient of variation, time in range in pregnancy 3.5-7.8 mmol/l, time above range in pregnancy >7.8 mmol/l and time below range in pregnancy <3.5 mmol/l between intervention and controls
Insulin and carbohydrates | Randomization, during pregnancy planning, study visits during pregnancy, around delivery and at one month post-delivery
  Total daily insulin dose, percentage insulin administered as basal insulin, carbohydrate-to-insulin ratio, numbers of boluses (automatic and manual), daily amount of entered carbohydrates
System features | From inclusion until one month post-delivery
  * Use of specific features as auto mode, "Ease-off" and "Boost" functions (intervention group)
  * Use of specific features as auto mode, night mode, fake carbohydrates (women in the control group using AID systems other than the CamAPS FX system)
HbA1c | Inclusion, last before pregnancy, at 9, 21, 33 and 35 weeks
  HbA1c before pregnancy and HbA1c levels during pregnancy.
Severe hypoglycemia | 2 years - if not becoming pregnant in the study period - until leaving the study
  The incidence of severe hypoglycemia in the year preceding pregnancy, during pregnancy and in the first one-month period post-delivery
Ketoacidosis | During pregnancy planning OR during pregnancy and post-delivery
  The prevalence of diabetic ketoacidosis (positive ketones in urine or serum, pH ≤7·30 and/or bicarbonate ≤18 mmol/l)
Weight | At inclusion until one month post-delivery OR leaving the study
  Maternal gestational weight gain and weight retention one month post-delivery OR Weight at randomization and last weight before pregnancy
Fetal overgrowth | At birth
  The prevalence of fetal overgrowth, defined as the offspring birth weight standard deviation score >90th percentile
Pregnancy complications | 9 months
  Prevalence of induced abortion, miscarriage, gestational hypertension, preeclampsia, need for maternal corticosteroid treatment for fetal lung maturation, early preterm delivery (before 34 completed weeks), preterm delivery (before 37 completed weeks), preterm pre-labour rupture of the membranes
Birth complications | From delivery until one month post-delivery
  Prevalence of shoulder dystocia, birth canal trauma, mode of delivery (vaginal delivery, instrumental delivery, planned cesarean section, emergency cesarean section), postpartum hemorrhage, maternal death
Neonatal morbidity | At delivery until one month post-delivery
  Neonatal hypoglycemia with plasma glucose <2.2 mmol/l two hours after birth, neonatal hypoglycemia requiring treatment with intravenous glucose, jaundice, respiratory distress, transient tachypnoea, duration of stay in neonatal intensive care unit, total number of admission days, cord blood pH, stillbirths, infant death within one month post-delivery
Major congenital malformations | From delivery until one month post-delivery
  ICD10 Q00-Q99 or requiring medical or surgical treatment
Infant growth | One month post-delivery
  Evaluated by weight standard deviation score and health evaluated as days with hospitalization during the first month of life after discharge in the neonatal period
Lactation | One month post-delivery
  The prevalence of lactation

CONTACTS AND LOCATIONS:
Locations (8):
- Denmark (8):
  - Department of Gynecology and Obstetrics, Aalborg University Hospital, Aalborg, Aalborg
  - Department of Gynecology and Obstetrics, Aarhus University Hospital, Aarhus, Aarhus N
  - Steno Diabetes Center Aarhus, Aarhus, Aarhus N
  - Steno Diabetes Center Nordjylland, Aalborg, Gistrup
  - Steno Diabetes Center Copenhagen, Copenhagen, Herlev
  - Department of Gynecology and Obstetrics, Odense University Hospital, Odense, Odense C
  - Steno Diabetes Center Odense, Odense University Hospital, Odense, Odense C
  - Center for Pregnant Women with Diabetes, Rigshospitalet, Copenhagen

IPD SHARING:
Plan to Share IPD: No
IPD will be shared if it is a requirement at our institution.